CLINICAL TRIAL: NCT00909831
Title: A Phase I Trial of Hydroxychloroquine in Combination With Temsirolimus in Patients With Refractory Solid Tumors
Brief Title: Hydroxychloroquine and Temsirolimus in Treating Patients With Metastatic Solid Tumors That Have Not Responded to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000643294; UPCC-08908; 807931; WYETH-C-UPCC-03809
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Hydroxychloroquine; temsirolimus; Microscopy, Electron; Chromatography, High Pressure Liquid; Immunologic Techniques; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: hydroxychloroquine
Drug: temsirolimus
Other: electron microscopy
Other: high performance liquid chromatography
Other: immunologic technique
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: pharmacological study
Procedure: autophagy inhibition therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as hydroxychloroquine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving hydroxychloroquine together with temsirolimus may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of hydroxychloroquine when given together with temsirolimus in treating patients with metastatic solid tumors that have not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of hydroxychloroquine (HCQ) in combination with temsirolimus (TEM) in patients with metastatic refractory solid tumors.

Secondary

* Describe the toxicity of this regimen in these patients.
* Measure the response rate in patients treated with this regimen.

Tertiary

* Establish a population pharmacokinetic (PK) model for HCQ and its metabolites in combination with TEM.
* Use the population PK model to estimate the exposure of HCQ in individual patients.
* Compare PK parameters for this regimen to data from published single agent studies.
* Measure the change in median number of autophagic vesicles/cell in peripheral blood mononuclear cells with TEM alone and with TEM and HCQ and correlate these changes with HCQ exposure.

OUTLINE: This is a dose-escalation study of hydroxychloroquine.

Patients receive temsirolimus IV over 30 minutes once a week beginning in week 1 and oral hydroxychloroquine twice daily beginning in week 2. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for pharmacokinetic and pharmacodynamic studies and measurement of autophagy inhibition. Samples are analyzed via HPLC and tandem mass spectrometry, immunoblotting assays, and electron microscopy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory solid tumor for which no curative standard therapy exists

  * Metastatic disease
* Treated brain metastases that have been stable ≥ 3 months allowed

  * At least 1 week since prior steroids

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2 times upper limit of normal (ULN)
* ALT and AST ≤ 5 times ULN
* Total bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious concurrent infection or medical illness that would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* No prior or other concurrent malignancy except for curatively treated carcinoma-in-situ at any site or basal cell carcinoma or squamous cell carcinoma of the skin

  * Patients who have been free of disease (any prior malignancy) for ≥ 5 years are eligible
* No porphyria
* No psoriasis, except well controlled psoriasis under the care of a specialist
* No previously documented macular degeneration or diabetic retinopathy
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Any number and type of prior anticancer therapies allowed
* No prior mTOR inhibitors
* At least 4 weeks since prior immunotherapy (i.e., aldesleukin, interferon, CTLA-4) or chemotherapy and recovered
* At least 2 weeks since prior oral targeted therapy and recovered
* At least 4 weeks since prior and no other concurrent investigational anticancer therapy (except for vaccines)
* No other concurrent therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent cytochrome P450 enzyme-inducing anticonvulsant drugs (i.e., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine)
* Concurrent non-enzyme inducing anticonvulsants, including felbamate, valproic acid, gabapentin, lamotrigine, tiagabine, topiramate, zonisamide, or levetiracetam allowed
* Concurrent hematologic growth factors (filgrastim [G-CSF], pegfilgrastim, epoetin alfa) allowed in patients with severe myelosuppression

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of hydroxychloroquine

SECONDARY OUTCOMES:
Response rate
Toxicity rate as assessed by NCI CTCAE v. 3.0
Pharmacokinetic and pharmacodynamic correlative endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States